CLINICAL TRIAL: NCT06563687
Title: Real-time Continuous Glucose Monitoring in Infants With Hypoxic-ischaemic Encephalopathy: a Pilot Randomized Controlled Trial
Brief Title: Continuous Glucose Monitoring in HIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Paolo Montaldo, Principal Investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SecondUNI84
Record Dates: First submitted 2024-08-14; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hypoxic Ischemic Encephalopathy of Newborn; Hyperglycemia; Hypoglycemia
Keywords: Continuous glucose monitoring; Neonatal hypoglycemia; Neonatal hyperglycemia
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Unblinded CGM (Experimental): CGM data will be "unblinded", with alarms on for hypo and hyperglycemia. CGM data will be used to support clinical management including blood glucose measurements and decision making. Changes in glucose and insulin infusion will be based primarily on the real-time CGM data but blood glucose concentrations will be checked in case of rapid changes in CGM data or before any treatment.
  Interventions: Device: Dexcom ONE+
- Blinded CGM (Other): CGM data will be blinded. Alarms for Hypo and hyperglycemia will be off. Glucose control will be monitored and managed according to standard clinical practice using intermittently sampled blood glucose concentrations.
  Interventions: Device: Dexcom ONE+

INTERVENTIONS:
Device: Dexcom ONE+ — In all the neonates recruited CGM sensor and transmitter will be placed soon after study enrollment. The sensors will be inserted in the lateral thigh and continuous measurements will be recorded for all the duration of therapeutic hypothermia.

SUMMARY:
The aim of the study is to examine whether the use of continuous glucose monitoring (CGM) to guide the clinical management of glycaemic control will result into an increased time in the target glucose concentration. To further examine the efficacy of using CGM the following secondary outcomes in the two groups were assessed: mean glucose values, glucose variability within individuals, percentage of time that glucose values are in hyperglycaemic or hypoglycaemic ranges.

Randomized controlled trial recruiting neonates (Birth weight >1.8kg, Gestation>36 weeks) with moderate or severe hypoxic ischemic encephalopathy (HIE) following perinatal asphyxia . Neonates will be randomly assigned (1:1) within 6 hours of birth to receive either the intervention with real-time CGM or standard care for 72 hours.

DETAILED DESCRIPTION:
Neonatal hypoglycaemia and hyperglycaemia are associated with brain injury and impaired neurodevelopment outcomes in neonates with HIE. Improving early glucose control is an important modifiable risk factor for outcomes in this population. Glycaemic monitoring is usually performed by capillary or central line sampling. However, over 30% of the episodes of abnormal glucose concentration are undetected, even with regular but intermittent sampling. CGM can allow earlier detection and prevention of exposure to extreme glucose concentrations.

Study design - This is a multicentre interventional, open-label, randomized controlled trial of CGM compared with standard clinical management (control).A total of 70 neonates (Birth weight >1.8kg, Gestation >36 weeks and aged <6hours) with moderate or severe HIE following perinatal asphyxia will be recruited within 6 hours of birth after informed parental consent. Neonates with major congenital malformations, inborn errors of metabolism, congenital infections, imminent death will be excluded.

Neonates will be randomly assigned (1:1) to receive either the intervention with real-time CGM for 72 hours or standard care using a randomization program (R package SRS: A Subject Randomization System). We will use the minimization method to control for severity and to achieve balance within recruiting centres. In all the neonates recruited Dexcom ONE+ CGM (Dexcom, San Diego, CA, USA) will be placed soon after study enrollment. The sensors will be inserted in the lateral thigh and continuous measurements will be recorded for 72 h. The CGM device will be calibrated using blood glucose values measured by point-of-care test. CGM calibrations will be performed at least twice a day. CGM data will be downloaded by using Dexcom Studio software on a dedicated computer.

In the standard care group, the CGM device will collect glucose data continuously, but the clinical team will be blinded to the data. These neonates will have their glucose control monitored and managed according to standard clinical practice using intermittently sampled blood glucose levels. In the intervention group the CGM data will be used to support clinical management including blood glucose measurements and decision making. Changes in glucose and insulin infusion will be based primarily on the real-time CGM data but blood glucose concentrations will be checked in case of rapid changes in CGM data.

Interventions to target glucose control will be guided by a protocol shared among the participating hospitals. As part of the study protocol, all the neonates will receive a continuous infusion of glucose 10% of 3-4 mg/kg/minute and total fluid intake starting at 50-60 ml/kg/day followed by titration depending on urine output, renal function, and management of glucose infusion rates.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight >1.8kg
* Gestation >35 weeks
* Aged <6hours
* Moderate or severe HIE following perinatal asphyxia

Exclusion Criteria:

* Major congenital malformations
* Inborn errors of metabolism,
* Congenital infections
* Imminent death

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
In range - time | 72 hours after birth
  Proportion of time that the sensor glucose values are in the target range (50 to 180 mg/dL) compared between the study groups

SECONDARY OUTCOMES:
Hypoglycemia | 72 hours after birth
  Percentage of time below 50 mg/dl
Hyperglycemia | 72 hours after birth
  Percentage of time above 180 mg/dl
Glycemic variability | 72 hours after birth
  Evaluation of glycemic variability
Adverse events associated to insertion of CGM | up to 10 days after birth
  % of infants with adverse events secondary to CGM placement or wear

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - A.O.S.G. Moscati, Avellino
  - Monaldi | | AORN - Ospedali dei ColliAORN - Ospedali dei Colli, Naples
  - University of Campania Luigi Vanvitelli, Napoli

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available when scientific manuscripts are published.
  Data that cannot be shared publicly (e.g. to protect patient confidentiality) will be by request only. The PI will review each request on case-by-case basis. Upon approval the data requester will be asked to sign a data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available 1 to 2 years after the end of the study.
Access Criteria: Unidentified data will be shared by publication. Request for data that affects patient confidentiality will review by the study PI on a case-by-case basis.

REFERENCES:
- [Background] Kalogeropoulou MS, Thomson L, Beardsall K. Continuous glucose monitoring during therapeutic hypothermia for hypoxic ischaemic encephalopathy: a feasibility study. Arch Dis Child Fetal Neonatal Ed. 2023 May;108(3):309-315. doi: 10.1136/archdischild-2022-324593. Epub 2022 Dec 20. PMID 36600516
- [Background] Pinchefsky EF, Hahn CD, Kamino D, Chau V, Brant R, Moore AM, Tam EWY. Hyperglycemia and Glucose Variability Are Associated with Worse Brain Function and Seizures in Neonatal Encephalopathy: A Prospective Cohort Study. J Pediatr. 2019 Jun;209:23-32. doi: 10.1016/j.jpeds.2019.02.027. Epub 2019 Apr 11. PMID 30982528
- [Background] Montaldo P, Caredda E, Pugliese U, Zanfardino A, Delehaye C, Inserra E, Capozzi L, Chello G, Capristo C, Miraglia Del Giudice E, Iafusco D. Continuous glucose monitoring profile during therapeutic hypothermia in encephalopathic infants with unfavorable outcome. Pediatr Res. 2020 Aug;88(2):218-224. doi: 10.1038/s41390-020-0827-4. Epub 2020 Mar 2. PMID 32120381
- [Background] Mietzsch U, Wood TR, Wu TW, Natarajan N, Glass HC, Gonzalez FF, Mayock DE, Comstock BA, Heagerty PJ, Juul SE, Wu YW; HEAL Study Group. Early Glycemic State and Outcomes of Neonates With Hypoxic-Ischemic Encephalopathy. Pediatrics. 2023 Oct 1;152(4):e2022060965. doi: 10.1542/peds.2022-060965. PMID 37655394
- [Background] Parmentier CEJ, de Vries LS, van der Aa NE, Eijsermans MJC, Harteman JC, Lequin MH, Swanenburg de Veye HFN, Koopman-Esseboom C, Groenendaal F. Hypoglycemia in Infants with Hypoxic-Ischemic Encephalopathy Is Associated with Additional Brain Injury and Worse Neurodevelopmental Outcome. J Pediatr. 2022 Jun;245:30-38.e1. doi: 10.1016/j.jpeds.2022.01.051. Epub 2022 Feb 2. PMID 35120986
- [Background] Basu SK, Kaiser JR, Guffey D, Minard CG, Guillet R, Gunn AJ; CoolCap Study Group. Hypoglycaemia and hyperglycaemia are associated with unfavourable outcome in infants with hypoxic ischaemic encephalopathy: a post hoc analysis of the CoolCap Study. Arch Dis Child Fetal Neonatal Ed. 2016 Mar;101(2):F149-55. doi: 10.1136/archdischild-2015-308733. Epub 2015 Aug 17. PMID 26283669
- [Background] Tam EWY, Kamino D, Shatil AS, Chau V, Moore AM, Brant R, Widjaja E. Hyperglycemia associated with acute brain injury in neonatal encephalopathy. Neuroimage Clin. 2021;32:102835. doi: 10.1016/j.nicl.2021.102835. Epub 2021 Sep 28. PMID 34601311
- [Background] Puzone S, Diplomatico M, Caredda E, Maietta A, Miraglia Del Giudice E, Montaldo P. Hypoglycaemia and hyperglycaemia in neonatal encephalopathy: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2023 Dec 15;109(1):18-25. doi: 10.1136/archdischild-2023-325592. PMID 37316160
- [Background] Kamino D, Widjaja E, Brant R, Ly LG, Mamak E, Chau V, Moore AM, Williams T, Tam EWY. Severity and duration of dysglycemia and brain injury among patients with neonatal encephalopathy. EClinicalMedicine. 2023 Mar 23;58:101914. doi: 10.1016/j.eclinm.2023.101914. eCollection 2023 Apr. PMID 37181414